CLINICAL TRIAL: NCT06996613
Title: Liberal Versus Restrictive Transfusion Strategy in Patients With Upper Git Bleeding in Sohag University Hospital
Brief Title: Liberal Versus Restrictive Transfusion Strategy in Patients With Upper Git Bleeding
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Elsayed Ibrahim, resident doctor, Sohag University
Other Study IDs: Soh-Med--25-5-12MS
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Upper Git Bleeding
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Upper endoscopy — It's a diagnostic endoscope to show the cause of upper Git bleeding

SUMMARY:
Comparison between the effects and results of the two strategies of blood transfusion, liberal and restrictive in patients with upper Git bleeding

DETAILED DESCRIPTION:
Comparison between safety, efficacy and mortality rate in the two strategies of blood transfusion, liberal(target Hb 9-11g/dl) and restrictive(target Hb 7-9 g/dl )in patients with upper Git bleeding in sohag university hospital, and how other risk factors as liver cirrhosis , CKD,and cause of bleeding in the patient affect results and expected complications that may be occur after blood transfusion

ELIGIBILITY:
Inclusion Criteria:

* all patients presented by upper GIT bleeding and their CBC show anemia and need blood transfusion

Exclusion Criteria:

* all patients less than 18 years and patients have anemia and received blood transfusion by another causes other than GIT bleeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper Git bleeding in sohag university hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-22 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
the rate of complication of both liberal and restrictive transfusion strategy in upper Git bleeding | Baseline
  To assess outcomes and any unwanted complications of both liberal and restrictive transfusion strategy in patients with upper GIT bleeding after reaching target Hb

CONTACTS AND LOCATIONS:
Overall Officials: Reham Elsayed, Study Chair — Sohg university hospital; Reham Elsayed, Principal Investigator — Tertiary hospital
Locations (1):
- Faculty of medicine sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Risk of re identification of participant data and privacy concerns
  * Reuse of data for proposes that had not been approved by participants
  * Reuse of data for unfair commercial proposes